CLINICAL TRIAL: NCT07245706
Title: Ensuring Shoulder Health as a Key Factor for Long Term Health and Functioning of Manual Wheelchair Users
Brief Title: Shoulder Health After Rehabilitation and Performance Training
Acronym: SHARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-16; 10.003.991 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2025-10-01; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Nervous System Diseases; Musculoskeletal Diseases; Injury
Keywords: Shoulder; Wheelchair; Training; Activity of Daily Life; Load; Capacity; Functioning; Monitoring
MeSH Terms: conditions — Spinal Cord Injuries; Nervous System Diseases; Musculoskeletal Diseases; Wounds and Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The general radiologist who assesses the MRI images will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Experimental): This group starts the training program 3 months post discharge from primary rehabilitation after spinal cord injury
  Interventions: Other: Strength training
- Late intervention (Experimental): This group starts the training program 12 months post discharge from primary rehabilitation after spinal cord injury
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — Individualized, home-based strength trainig consisting of 6 ecxercises that will be carried out twice a week for 12 weeks

SUMMARY:
The goal of this study is to investigate the impact of a home-based shoulder strength training on the overall shoulder health in manual wheelchair users, and if the timepoint of such a training makes a difference. The study is focusing on persons with a spinal cord injury in the thoracic or lumbar region of the spine, that have only recently been injured and will soon be discharged from primary rehabilitation.

The shoulder training will take place either 3 or 12 months after discharge from primary rehabilitation and will be carried out twice a week for 12 weeks.

There are six measurements occurring every three months, which leads to an overall duration of 15 months. The measurements consist of:

* Questionnaires about independence in daily life, participation, quality of life and physical activity
* Assessment of shoulder strength, range of motion and function
* Measurement of the daily wheelchair use during one week via sensors that are fixed to the wheelchair and wrist
* one further questionnaire at the end of the measurement week about the occurrence of shoulder pain

Additionally, on four of the six measurement timepoints, a magnet resonance image (MRI) of the shoulder will be taken to assess the shoulder status (pathology, muscle volume and quality).

Though all these measurements the researchers can additionally assess the load of daily life on the shoulders, and how well this matches the preparation during the primary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a paraplegia below T2
* Manual wheelchair user
* Age 18 - 70 years
* At discharge from initial rehabilitation

Exclusion Criteria:

* Trauma or surgery of the shoulder with medical indication for immobilization of more than four weeks
* Constant use of power assistance for the wheelchair
* Any surgical implants that exclude the participant for MRI assessments of the shoulder
* Inability to follow the study instructions, e.g., mental health problems, language problems, dementia, claustrophobia (for MRI) etc.
* Persons with congenital conditions leading to SCI, SCI in the context of palliative care, neurodegenerative disorders, and Guillain-Barré syndrome
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
change in experienced shoulder pain during activities of daily life | Before and after the training intervention (3 months apart)
  Expressed by the Wheelchair User's Shoulder Pain Index (WUSPI) score, a validated 15-item self-report instrument measuring shoulder pain during activities of daily life. For each activity, the shoulder pain experienced during the preceding week (corresponding to the week of monitoring of external exposure) is scored using a Visual Analog Scale (0-10). Total index scores can range from zero to 150 with zero meaning no pain and 150 maximal possible pain.

SECONDARY OUTCOMES:
Experienced shoulder pain during activities of daily life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Expressed by the Wheelchair User's Shoulder Pain Index (WUSPI) score, a validated 15-item self-report instrument measuring shoulder pain during activities of daily life. For each activity, the shoulder pain experienced during the preceding week (corresponding to the week of monitoring of external exposure) is scored using a Visual Analog Scale (0-10). Total index scores can range from zero to 150 with zero meaning no pain and 150 maximal possible pain.
Painful events | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Specific events that resulted in shoulder pain during the measurement week
Shoulder strength | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  excerted peak force during six shoulder movements (abduction, adduction, flexion, extension, internal rotation, and external rotation), measured with a force sensor
Shoulder range of motion | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  active and passive range of motion of six shoulder movements (abduction, adduction, flexion, extension, internal rotation, and external rotation), measured with a goniometer
Shoulder stability | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Assessed with clinical tests (provocative testing); Aggregated tests against resistance in eight different positions:
  * Full can test
  * Empty can test
  * Gerber's Lift off test
  * Neer's Test
  * Hawkins-Kennedy Test
  * Yergason's Test
  * Crank's Test
  * Belly-Press Test
  Rated as painful, weak, negative, or not possible
Heart rate during daily life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  variation over the day, assessed by a wrist sensor
Wheelchair use during daily life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge, measured for one week each
  Quantified by characteristics such as distance covered, number of pushes and turns or propulsion on an incline, measured by inertial measurement units (IMUs)
Shoulder loading acivities of daily life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge, measured for one week each
  Classified by a machine learning algorithm including wheelchair propulsion, weight relief lift, manual material handling, transfer and deskwork, measured by inertial measurement units (IMUs) and a wheelchair cushion pressure mat
Shoulder load during activities of daily life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge, measured for one week each
  Total shoulder load calculated based on the frequency and duration of the activities and the shoulder load related to these activities
Shoulder pathology | 3, 6, 12 and 15 months after discharge
  Grading of MRI abnormalities of rotator cuff tendons including tendinopathy and tendon tears and determination of Total Tendon Score (range 0-40)
Shoulder muscle volume | 3, 6, 12 and 15 months after discharge
  Quantification of the muscle volume of the rotator cuff by deep-learning-based segmentation of the MRI
Shoulder muscle quality | 3, 6, 12 and 15 months after discharge
  Quantification of fatty infiltration (fat fraction) of the rotator cuff by deep-learning-based segmentation of the MRI
Independence during daily life | 3, 6, 12 and 15 months after discharge
  Quantified by the Self Report Spinal Cord Independence Measure (SR-SCIM)., a valid 17-item self-report instrument measuring independence in the domains of self-care, respiration and sphincter management and mobility. Total index scores can range from zero to 100.
Participation | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Assessed with the Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P), a valid 31-item instrument measuring participation in the domains of frequency, restrictions and satisfaction
General quality of life | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Quantified by the 12-Item Short Form Survey (SF-12), a self-reported outcome measure assessing the impact of health on an individual's everyday life. Total scores can range from zero to 100
Physical activity | Before discharge from primary rehabilitation, 3, 6, 9, 12 and 15 months past discharge
  Assessed by the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD), a 13-item questionnaire assessing physical activity over the preceding week in the domains of leisure, household and occupational activity. Scores are quantified in Metabolic Equivalents (METS h/day) and range from 0 (no activity) to over 100 METS h/day (very high)

OTHER OUTCOMES:
Training amount | During the 12 weeks training intervention, after each session
  Number of repetitions of each exercise of the shoulder training will be recorded via the PhysiApp
Training resistance | During the 12 weeks training intervention, after each session
  Resistance used (e.g. weight) during the shoulder training will be recorded via the PhysiApp
Training exhaustion | During the 12 weeks training intervention, after each session
  Exhaustion felt during the shoulder training will be recorded via the PhysiApp on a scale from one to ten, where ten is highest exhaustion possible

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No